CLINICAL TRIAL: NCT05773560
Title: Investigation of the Influence of Virtual Reality on the Postoperative Period After Major Amputation.
Brief Title: Virtual Reality in the Rehabilitation in Patients With Lower Limb Amputation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Ulrich Rother, PD Dr. med., University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VR-amputation
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Amputation; Lower Limb; Rehabilitation; Activities of Daily Living; Virtual Reality; Lower Extremity
Keywords: Amputation; Lower Extremity Ischemia; Lower Limb; Lower Limb Ischemia; Rehabilitation; Activities of Daily Living; Virtual Reality; Lower Limb Amputation Knee; Lower Limb Amputation Above Knee; Lower Limb Amputation Below Knee; Lower Extremity Wound

STUDY DESIGN:
Intervention Model Description: Patients after a major amputation would received at least 10 days of rehabilitation with the assistance of virtual reality. Before the operation, patients consent, life quality, pain score and motivation score were be evaluated. The rehabilitation with virtual reality started on the second postoperative day. The pain score would be evaluated everyday before and after the rehabilitation. On the fifth and tenth day, motivation, life quality and functional index would be carried out again as the evaluation of the outcome of training.
Masking Description: The researcher analyzing the final outcomes is blinded from the personal information and execution of the rehabilitation of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving rehabilitation with virtual reality. (Experimental): Single Group Assignment Patients after a major amputation would received at least 10 days of rehabilitation with the assistance of virtual reality. Before the operation, patients consent, life quality, pain score and motivation score were be evaluated. The rehabiliation with virtual reality started on the second postoperative day. The pain score would be evaluated everyday before and after the rebilitation. On the fifth and tenth day, motivation, life quality and functional index would be carried out again as the evaluation of the outcome of training.
  Interventions: Device: virtual reality rehabilitation

INTERVENTIONS:
Device: virtual reality rehabilitation — All patients will receive VR-assisted rehabilitation. The VR-assisted rehabilitation is proceed with SyncVR® (Padualaan, Netherlands ) equipment, which is composed of a head set (PICO NEO 3) and one dashboard (TABLET), enabling the patients to receive stepwise rehabilitation program with 360° videos activities (SyncVR Medical Platform). The VR-assisted rehabilitation will be performed two times per day, 30 minutes per training. The first training will start on the second post-operative day.

SUMMARY:
The goal of this clinical trial is to test the impact of virtual reality on rehabilitation for the patients after a major amputation.

The main questions it aims to answer are:

* Does the virtual-reality-assisted rehabilitation improve the life quality of patients (i.e. lesser pain, better spirit)?
* Does the virtual-reality-assisted rehabilitation improve the daily life function of the patients? Participants will received a virtual-reality-assisted rehabilitation on the second postoperative day for ten days. The rehabilitation would be carried out two times per day and 30 minutes per training.

DETAILED DESCRIPTION:
Despite the increasing development of revascularisation techniques, lower limb amputation often represent the last chance of survival for the vasculopathic patient with chronic limb threatening ischemia (CLTI). First goal after lower limb amputation is represented by a rapid prosthesis application. The patient in the immediate post-operative period must undergo intensive rehabilitation and physiotherapy, which involves not only a physical but also a psychological approach.

"Classical" recovery following lower limb amputation includes adequate pain therapy and physiotherapy to regain independence, strength, mobility and finally prothesis application to improve quality of life and restore mobility. The aim of this study is to investigate the effect of adding virtual reality to traditional rehabilitation following a lower limb amputation in patients due to limited circulation, with particularly attention to a possible improvement of psychological state, reduction of post-operative pain and more rapid improvement in regaining functional mobility

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* critical limb ischemia or acute limb ischemia
* amputation above/below knee
* unilateral lower limb amputees

Exclusion Criteria:

* physical disability (paralysis, plegia)
* inability to give informed consent
* neurological or psychiatric problem that reduces compliance
* loss of planned post-operative assessments
* traumatic amputation in a patient without circulatory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | single time point (1 day)
  The change in activities of daily life among the patients before and after the implementation of the training program.
The Morton Mobility Index (DEMMI) | single time point (1 day)
  The change in mobility outcomes among the patients before and after the implementation of the training program.
Esslinger Transfer Scale | single time point (1 day)
  The change in the level of assistance needed for a safe transfer among the patients before and after the implementation of the training program.

SECONDARY OUTCOMES:
SF-12® Health Survey | single time point (1 day)
  The change in life quality in terms of both mentally and physically among the patients before and after the implementation of the training program.
6-point Likert-scale | single time point (1 day)
  The change in pain among the patients before and after the implementation of the training program.
Situational Motivational Scale | single time point (1 day)
  The change in motivation among the patients before and after the implementation of the training program.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen-Nuremberg (FAU), Department of Vascular Surgery, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Esquenazi A. Amputation rehabilitation and prosthetic restoration. From surgery to community reintegration. Disabil Rehabil. 2004 Jul 22-Aug 5;26(14-15):831-6. doi: 10.1080/09638280410001708850. PMID 15497912
- [Background] Rau B, Bonvin F, de Bie R. Short-term effect of physiotherapy rehabilitation on functional performance of lower limb amputees. Prosthet Orthot Int. 2007 Sep;31(3):258-70. doi: 10.1080/03093640600994615. PMID 17979011
- [Background] Andrysek J, Klejman S, Steinnagel B, Torres-Moreno R, Zabjek KF, Salbach NM, Moody K. Preliminary evaluation of a commercially available videogame system as an adjunct therapeutic intervention for improving balance among children and adolescents with lower limb amputations. Arch Phys Med Rehabil. 2012 Feb;93(2):358-66. doi: 10.1016/j.apmr.2011.08.031. PMID 22289250
- [Background] Murray CD, Patchick E, Pettifer S, Caillette F, Howard T. Immersive virtual reality as a rehabilitative technology for phantom limb experience: a protocol. Cyberpsychol Behav. 2006 Apr;9(2):167-70. doi: 10.1089/cpb.2006.9.167. PMID 16640472
- [Background] Rothgangel A, Bekrater-Bodmann R. Mirror therapy versus augmented/virtual reality applications: towards a tailored mechanism-based treatment for phantom limb pain. Pain Manag. 2019 Mar 1;9(2):151-159. doi: 10.2217/pmt-2018-0066. Epub 2019 Jan 25. PMID 30681034
- [Background] de Rooij IJM, van de Port IGL, Punt M, Abbink-van Moorsel PJM, Kortsmit M, van Eijk RPA, Visser-Meily JMA, Meijer JG. Effect of Virtual Reality Gait Training on Participation in Survivors of Subacute Stroke: A Randomized Controlled Trial. Phys Ther. 2021 May 4;101(5):pzab051. doi: 10.1093/ptj/pzab051. PMID 33594443
- [Background] Dominguez-Navarro F, Igual-Camacho C, Silvestre-Munoz A, Roig-Casasus S, Blasco JM. Effects of balance and proprioceptive training on total hip and knee replacement rehabilitation: A systematic review and meta-analysis. Gait Posture. 2018 May;62:68-74. doi: 10.1016/j.gaitpost.2018.03.003. Epub 2018 Mar 5. PMID 29525292
- [Background] Smits M, Staal JB, van Goor H. Could Virtual Reality play a role in the rehabilitation after COVID-19 infection? BMJ Open Sport Exerc Med. 2020 Oct 23;6(1):e000943. doi: 10.1136/bmjsem-2020-000943. eCollection 2020. PMID 33178449
- [Background] de Morton NA, Davidson M, Keating JL. The de Morton Mobility Index (DEMMI): an essential health index for an ageing world. Health Qual Life Outcomes. 2008 Aug 19;6:63. doi: 10.1186/1477-7525-6-63. PMID 18713451